CLINICAL TRIAL: NCT03606057
Title: A Randomized, Double-Blind, Parallel, Nested Crossover Study to Investigate the Effect of JNJ-64565111 on Cardiac Repolarization (Corrected QT Interval) Compared With Placebo in Healthy Adults: a Thorough ECG Study Employing Placebo, JNJ-64565111, and a Positive Control (Moxifloxacin)
Brief Title: A Study to Investigate the Effect of JNJ-64565111 on Cardiac Repolarization (Corrected QT Interval) Compared With Placebo in Healthy Adults: a Thorough ECG Study Employing Placebo, JNJ-64565111, and a Positive Control (Moxifloxacin)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108477; 64565111OBE1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-07-10; First posted 2018-07-30 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1: JNJ-64565111+Moxifloxacin Placebo (Experimental): Participant will receive JNJ-64565111 on days 2, 9, 16, and 23 and moxifloxacin-matching placebo on days 1 and 27.
  Interventions: Drug: JNJ-64565111; Drug: Moxifloxacin-matching Placebo
- Treatment Group 2: JNJ-64565111 Matching Placebo+Moxifloxacin (Active Comparator): Participant will receive JNJ-64565111-matching placebo on days 2, 9, 16, and 23. Participants will also receive moxifloxacin on day 1 and moxifloxacin-matching placebo on day 27 (sequence 2a) or moxifloxacin-matching placebo on day 1 and moxifloxacin on day 27 (sequence 2b) in a nested crossover manner.
  Interventions: Drug: Moxifloxacin; Drug: JNJ-64565111-matching Placebo; Drug: Moxifloxacin-matching Placebo

INTERVENTIONS:
Drug: JNJ-64565111 — Participants will receive JNJ-64565111, subcutaneously on days 2, 9, 16, and 23.
  Arms: Treatment Group 1: JNJ-64565111+Moxifloxacin Placebo
Drug: Moxifloxacin — Participants will receive moxifloxacin capsule on days 1 or 27 in a nested crossover manner.
  Arms: Treatment Group 2: JNJ-64565111 Matching Placebo+Moxifloxacin
Drug: JNJ-64565111-matching Placebo — Participants will receive JNJ-64565111-matching Placebo vehicle solution subcutaneously on days 2, 9, 16, and 23.
  Arms: Treatment Group 2: JNJ-64565111 Matching Placebo+Moxifloxacin
Drug: Moxifloxacin-matching Placebo — Participants will receive moxifloxacin-matching placebo capsule on days 1 and 27 in treatment group 1 and on day 1 or 27 in treatment group 2.

SUMMARY:
The purpose of this study is to assess the effects on placebo-corrected change from baseline QT interval corrected for individual heart rate (QTcI) of JNJ-64565111 close to steady state on Day 26 and on electrocardiogram morphology at supratherapeutic exposures in otherwise healthy overweight/obese adults after 4 weeks of treatment with JNJ 64565111 administered subcutaneously once weekly.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25.0 and 40.0 kilogram per square meter ( kg/m^2), inclusive, and a body weight of not less than 80 kg
* Blood pressure (BP) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* If a woman, must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study (from screening through Day 56) or until 30 days after the last dose of study drug for participants that withdraw early from the study
* QRS interval of less than or equal to (<=) 110 milliseconds (ms)
* An average of triplicate 12-lead safety electrocardiogram (ECG) recording, completed within 4 minutes total, consistent with normal cardiac conduction and function at screening, including

  1. Normal sinus rhythm (heart rate between 45 and 100 beats per minute [inclusive])
  2. QT interval corrected for heart rate according to Fridericia's formula (QTcF) interval between 350 to 450 ms (inclusive)
  3. PR interval <= 200 ms
  4. ECG morphology consistent with healthy cardiac conduction and function

Exclusion Criteria:

* Taken any disallowed therapies as defined in a protocol before the planned first dose of study drug
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram at screening or at admission to the study site
* Known allergies, hypersensitivity, or intolerance to JNJ-64565111, moxifloxacin, or its excipients
* Hepatitis B or C infection
* History of additional risk factors for torsade de pointes or the presence of a family history of Short QT Syndrome, Long QT Syndrome, sudden unexplained death at a young age (<= 40 years), or sudden infant death syndrome in a first-degree relative (that is biological parent, sibling, or child)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Placebo-Corrected Change from Baseline in QT Interval Corrected for Individual Heart Rate (QTcI) on Day 26 Time-Matched Time Points | Baseline and Day 26
  Placebo-corrected change from baseline in QT interval corrected for individual heart rate (QTcI) on day 26 time-matched time points will be determined. The mean change from baseline in QTcI for participants who receive placebo will be subtracted from the mean change from baseline in QTcI for participants on JNJ-64565111 at the same time point to generate placebo-corrected change from baseline in QTcI, which will be presented.
Change from Time-Matched Baseline in QTc Interval | Up to Day 27
  The QT interval corrected for heart rate (QTc interval) using Fridericia method will be measured by electrocardiograms (ECG).
Change from Time-Matched Baseline in Heart Rate (HR) | Up to Day 27
  The HR will be measured by ECG.
Change from Time-Matched Baseline in QRS Interval | Up to Day 27
  The QRS Intervals will be measured by ECG.
Change from Time-Matched Baseline in PR Interval | Up to Day 27
  The PR intervals will be measured by ECG.

SECONDARY OUTCOMES:
Cardiac Repolarization as Determined by Mean Change from Time-Matched Baseline in QT Interval Corrected for Individual HR (QTcI) on Day 5 | Baseline and Day 5
  Mean change from time-matched baseline in QT interval corrected for individual HR (QTcI) on day 5 to determine the effect of JNJ-64565111 on cardiac repolarization.
Cardiac Repolarization as Determined by Mean Change from Time-Matched Baseline in QT Interval Corrected For HR Using Fridericia's Formula (QTcF) on Day 5 and Day 26 | Baseline, Day 5 and Day 26
  Mean change from time-matched baseline in QT interval corrected for HR using Fridericia's formula (QTcF) will be assessed on day 5 and day 26 to determine the effect of JNJ-64565111 on cardiac repolarization.
Maximum Observed Serum Concentration (Cmax) | Days 1, 5, 26 and 27
  Cmax is defined as the maximum observed serum analyte concentration.
Time to Reach Maximum Observed Serum Concentration (Tmax) | Days 1, 5, 26 and 27
  Tmax is defined as actual sampling time to reach maximum observed serum analyte concentration.
Average Serum Analyte Concentration (Cavg) | Days 1, 5, 26 and 27
  Cavg is defined as average serum analyte concentration.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From signing of the informed consent form (ICF) to end of study (approximately 12 weeks)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
QTcI Changes Evaluated Using ECG Assessments versus Serum Concentrations of JNJ-64565111 | Up to Day 27
  QTcI changes evaluated using ECG assessments versus serum concentrations of JNJ-64565111 will be quantified. QTcI is a QT interval corrected for heart rate using individual-specific correction formula and QTcI changes will be quantified using a linear or nonlinear mixed effects modeling approach.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States